CLINICAL TRIAL: NCT05825976
Title: The Influence of Omega-3 Fatty Acid Supplementation on The Tear Film Quality in Celiac Patients
Brief Title: Omega-3 Fatty Acid Supplementation and Tear Film Quality in Celiac Patients
Acronym: OmegaCelDED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: Plava Medical Group, Bosna and Herzegovina (Unknown)
Responsible Party: Principal Investigator, Ines Banjari, Associate Professor, Clinical Nutrition Specialist, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBanjari
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye Syndromes; Celiac Disease
Keywords: Celiac Disease; Supplementation; Omega-3 Fatty Acids; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes; Celiac Disease | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Supplementation with 2 gel-capsules (each containing 720 mg eicosapentaenoic acid (EPA) and 480 mg docosahexaenoic acid (DHA))
  Interventions: Dietary Supplement: Omega-3 Fatty ACids
- Intervention group 2 (Experimental): Supplementation with 2 gel-capsules (each containing 320 mg eicosapentaenoic acid (EPA) and 200 mg docosahexaenoic acid (DHA))
  Interventions: Dietary Supplement: Omega-3 Fatty ACids
- Control (Active Comparator): Supplementation with 2 gel-capsules (each containing 1000 mg extra virgin olive oil)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty ACids — Intervention consists of two different doses of omega-3: high concentration (Intervention group 1) and low concentration (Intervention group 2).
  Arms: Intervention group 1; Intervention group 2
Other: Control — Supplementation with extra virgin olive oil as a for of positive placebo control.
  Arms: Control

SUMMARY:
The study aims to determine the effectiveness on the tear film quality and symptoms related with dry eye disease in patients with celiac disease.

DETAILED DESCRIPTION:
Patients diagnosed with celiac disease will be recruited for the study. They will be randomly assigned to one of the three arms (Intervention group 1 - high dose EPA and DHA, Intervention group 2 - low dose EPA and DHA, or Control - extra virgin olive oil) and for 45 days take supplementation as instructed. During the intervention they will be instructed to maintain their diet and lifestyle (i.e. they will not receive any education on diet or lifestyle modification). At inclusion, patients will complete one basic questionnaire on sociodemographic data, one questionnaire which assess accidental exposure to gluten and their weight and height will be measured. Subjective symptoms related to dry eye disease will be assessed with Ocular Surface Disease Index (OSDI) test, while quality and quantity of the tear film will be assessed with the Schirmer's test I and Tear Break-up Time test (TBUT). Dietary intake of omega-3 acids will be controlled by one 24-hour dietary recall (completed at inclusion an after the intervention).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of celiac disease
* signed informed consent form

Exclusion Criteria:

* use of medications for diabetes, hypertension, depression, thyroid disease, allergies, epilepsy, psychosis, glaucoma
* use of oral contraceptive pills
* alcoholism or use of alcohol on the day of recruitment
* menopause
* eye trauma or surgery in the past 3 months
* wearing contact lens
* supplementation with omega-3 fatty acids regardless of the dose used in the past month
* not understanding Bosnian letter or language
* Informed consent form not signed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Subjective symptoms of Dry Eye | 45 days
  Ocular Surface Disease Index or OSID is a 12-item questionnaire which assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Each question is graded on a scale of 0 to 4, where 0 indicates none of the time; 1, some of the time; 2, half of the time; 3, most of the time; and 4, all of the time. The total OSDI score is calculated as OSDI=[(sum of scores for all questions answered) × 100]/[(total number of questions answered) × 4]. Total score ranges from 0 to 100 where higher score coresponds with greater disability.
Tear Break-up Time | 45 days
  Used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film, as seen in this progression of these slit lamps photos over time. A TBUT under 10 seconds is considered abnormal.
Schirmer tear test | 45 days
  Evaluates aqueous tear production and is helpful in the assessment of patients with signs and/or symptoms of dry eye. Interpretation: normal aqueous tear production is supported by measurements of > 15 mm after 5 minutes, and mild-moderate reduction of aqueous production: 5mm-14mm after 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ines Banjari, PhD, Principal Investigator — Josip Juraj Strossmayer University of Osijek, Faculty of Food Technology, Department of Food and Nutrition Research
Locations (1):
- Plava Medical Group, Tuzla, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No
This research is part of PhD project and therefore the results cannot be shared directly. All interested parties can contact investigators after defending the PhD thesis.